CLINICAL TRIAL: NCT02236767
Title: Transcranial Magnetic Stimulation Treatment of Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIEF003523.4
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Hoarding
MeSH Terms: conditions — Hoarding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rTMS Treatment (Experimental): NeuroStar Transcranial Magnetic Stimulation Therapy System
  Interventions: Device: Neurostar Transcranial Magnetic Stimulation Therapy System

INTERVENTIONS:
Device: Neurostar Transcranial Magnetic Stimulation Therapy System — Treatment will entail daily (5 days/week) sessions of repetitive transcranial magnetic stimulation for 6 weeks employing right-sided, low frequency stimulation (1 Hz, 900 pulses/session for 30 sessions, 27,000 total pulses, intensity at 90% of the passive motor threshold) to the dorsolateral prefrontal cortex (DLPFC).

SUMMARY:
This is multiple baseline study including up to three participants with a primary diagnosis of hoarding disorder. All patients will receive unblinded repetitive transcranial magnetic stimulation study intervention.

DETAILED DESCRIPTION:
Study assessments will be conducted at pre-baseline, weekly during baseline assessment (until a stable baseline is established, but not less than 2, 4, and 6 weeks for patients respectively), weekly during treatment, and at post-treatment. Magnetic resonance imaging (MRI) will be competed at pre-baseline, pre-treatment, and post-treatment. Treatment will entail daily (5 days/week) sessions of repetitive transcranial magnetic stimulation using the Neurostar Therapy System for 6 weeks employing right-sided, low frequency stimulation (1 Hz, 900 pulses/session for 30 sessions, 27,000 total pulses, intensity at 90% of the passive motor threshold) to the dorsolateral prefrontal cortex (DLPFC). Neuronavigation will direct coil placement over the DLPFC based upon structural MRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hoarding disorder as primary disorder
* Clinical Global Impression Score > 3
* Saving Inventory-Revised score > 39

Exclusion Criteria:

* Any contraindication for participation in magnetic resonance imaging or transcranial magnetic stimulation
* Severe and/or unstable medical or psychiatric condition that require immediate medical attention
* Diagnosed with current major depressive episode
* Currently taking psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen J Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diefenbach GJ, Tolin DF, Hallion LS, Zertuche L, Rabany L, Goethe JW, Assaf M. A case study of clinical and neuroimaging outcomes following repetitive transcranial magnetic stimulation for hoarding disorder. Am J Psychiatry. 2015 Nov 1;172(11):1160-2. doi: 10.1176/appi.ajp.2015.15050602. No abstract available. PMID 26575452

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Therapy: NeuroStar TMS Therapy System
  Neurostar TMS Therapy System: Treatment will entail daily (5 days/week) sessions of rTMS for 6 weeks employing right-sided, low frequency stimulation (1 Hz, 900 pulses/session for 30 sessions, 27,000 total pulses, intensity at 90% of the passive motor threshold) to the dorsolateral prefrontal cortex (DLPFC).
Period: Overall Study
Arm/Group | TMS Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TMS Therapy
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Saving Inventory-Revised (SI-R) Total Score
Description: The Saving Inventory-Revised (SI-R) is a self-report measure which includes 23 items assessing the severity of hoarding symptoms including difficulty discarding, acquiring, and clutter. The 23 items are added for a total score which ranges from 0 to 92 and with higher score indicating more severe hoarding symptoms.
Time Frame: Pre-baseline, Post-baseline/Pre-treatment, Post-treatment, 2-Month Follow-up
Measure: Number; unit: units on a scale
Groups:
- rTMS Treatment: NeuroStar TMS Therapy System
  Neurostar TMS Therapy System: Treatment will entail daily (5 days/week) sessions of rTMS for 6 weeks employing right-sided, low frequency stimulation (1 Hz, 900 pulses/session for 30 sessions, 27,000 total pulses, intensity at 90% of the passive motor threshold) to the dorsolateral prefrontal cortex (DLPFC).
Arm/Group | rTMS Treatment
Number analyzed (Participants) | 1
units on a scale
  Pre-baselne | 66
  Post-baseline/Pre-treatment | 60
  Post-treatment | 46
  2-Month Follow-up | 45

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: an adverse events checklist was administered
Arm/Group | TMS Therapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Therapy (N=1)
tapping sound (Surgical and medical procedures) | 1 (1)
pin prick sensation at treatment site (Skin and subcutaneous tissue disorders) | 1 (1)
pain discomfort at the treatment site (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
eye twitch (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No